CLINICAL TRIAL: NCT00473408
Title: The Effect of Radiotherapy and Temozolomide on the Tumor Vasculature and Stem Cells in Human High-grade Astrocytomas
Acronym: Gliomstudien
Status: Terminated | Type: Observational
Why Stopped: Moved to another country, not possible to recruit from abroad.
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, Hans Petter Eikesdal, MD PhD, Haukeland University Hospital
Other Study IDs: 15437; REK ID: 202.06 (Registry Identifier: Regional Ethics Committee)
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Anaplastic Astrocytoma; Glioblastoma Multiforme; Tumor Angiogenesis
Keywords: Glioma; DCE-MRI; Angiogenesis; Cancer stem cells; Tumor vasculature
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Glioma | interventions — Magnetic Resonance Imaging; Dynamic Contrast Enhanced Magnetic Resonance Imaging; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples and blood samples are collected and frozen for future analysis for tumor vascularization and tumor stem cells.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Functional MRI (DCE-MRI) — MRI examination with i.v. gadolinium contrast to assess blood perfusion in remaining tumor tissue.
Procedure: Blood sample — See protocol.
Procedure: Tumor sample — See protocol.

SUMMARY:
The purpose of the current trial is to explore whether the standard treatment with radiotherapy and temozolomide affect the tumor vasculature in patients with high-grade astrocytomas. If vascular effects are identified, future clinical trials can be proposed wherein anti-angiogenic agents are added to increase patient survival.

DETAILED DESCRIPTION:
Today's standard treatment with radiotherapy and temozolomide yields a life expectancy of 1.5-3 years in patients with high-grade astrocytomas. Thus, there is a need for further therapeutic improvements in this patient population. The purpose of the current trial is to explore whether radiotherapy and temozolomide affect the tumor vasculature in patients with high-grade astrocytomas. If vascular effects are identified, future clinical trials can be proposed wherein anti-angiogenic agents are added to increase patient survival. Additionally, stem cells within malignant brain tumors is an important new area of research in this patient population, and investigations herein could contribute to identify new predictive markers and therapeutic targets.

Primary objective: To assess the vascular perfusion and permeability characteristics of high-grade astrocytomas (anaplastic astrocytoma and glioblastoma multiforme) using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) in patients receiving radiotherapy and temozolomide. Furthermore to assess whether therapy-induced changes in tumor perfusion is correlated with progression-free survival.

Secondary objectives:

* Analyze circulating endothelial cells in the blood by flow cytometry to explore whether these cells can be used as an indirect estimate of angiogenesis in high-grade astrocytomas
* Analyze tumor specimens from patients that have had their gliomas debulked before commencing therapy

  * immunostaining of the tumor vasculature to assess microvessel density
  * immunostaining for tumor stem cells
  * flow cytometric assessment of dissolved tumor tissue to look for tumor stem cells
* Assess progression-free survival of all patients included in the study, in order to correlate the survival data with the above tissue sampling results.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary high-grade astrocytoma, i.e. anaplastic astrocytoma or glioblastoma multiforme.
* Have a WHO performance status 0-2 and be able to undergo outpatient treatment.
* Age ≥18 years.
* No pregnant or lactating patients can be included.
* Patients must have radiographically documented measurable disease postoperatively. At least one tumor lesion must be unidimensionally measurable as follows:

  * Tumor lesion > 10 mm on conventional MRI scan, T1-weighted series, after intravenous (i.v.) gadolinium chelate contrast.
* All diagnostic radiology studies must be performed within 28 days prior to registration.
* Absence of conditions making MRI scans impossible;

  * Cardiac pacemaker
  * Other ferromagnetic metal implants not authorised for use in MRI such as some types of cerebral aneurysm clips
  * Serious claustrophobia
  * Obesity (> 300 lb., 140 Kg)
* Patients who are receiving corticosteroids have to receive stable or decreasing doses for at least 14 days before entering the trial.
* No prior chemotherapy for high-grade astrocytoma
* Absence of opportunistic infections making temozolomide contraindicated.
* Minimum required laboratory data:

  * Hematology:

    * Absolute granulocytes > 1.0 x 10^9/L
    * Platelets > 100 x 10^9/L
  * Biochemistry:

    * Bilirubin < 1.5 x upper normal limit
    * INR < 1.5
    * Serum creatinine <1.5 x upper normal limit
* Adequate cognitive function in order to give informed consent.
* Absence of any psychological, familial or sociological condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given according to national and local regulations.

Exclusion Criteria:

* Lack of fulfillment of inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older diagnosed and operated for high-grade astrocytoma.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Petter Eikesdal, MD PhD, Principal Investigator — Institute of Biomedicine, University of Bergen, Jonas Lies vei 91, 5009 Bergen, Norway
Locations (1):
- Dept. of Oncology & Dept. of Radiology, Haukeland University Hospital, Bergen, Norway, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No
Only one patient was included before the study was terminated.

REFERENCES:
- [Background] Cao Y, Sundgren PC, Tsien CI, Chenevert TT, Junck L. Physiologic and metabolic magnetic resonance imaging in gliomas. J Clin Oncol. 2006 Mar 10;24(8):1228-35. doi: 10.1200/JCO.2005.04.7233. PMID 16525177
- [Background] Morgan B, Thomas AL, Drevs J, Hennig J, Buchert M, Jivan A, Horsfield MA, Mross K, Ball HA, Lee L, Mietlowski W, Fuxuis S, Unger C, O'Byrne K, Henry A, Cherryman GR, Laurent D, Dugan M, Marme D, Steward WP. Dynamic contrast-enhanced magnetic resonance imaging as a biomarker for the pharmacological response of PTK787/ZK 222584, an inhibitor of the vascular endothelial growth factor receptor tyrosine kinases, in patients with advanced colorectal cancer and liver metastases: results from two phase I studies. J Clin Oncol. 2003 Nov 1;21(21):3955-64. doi: 10.1200/JCO.2003.08.092. Epub 2003 Sep 29. PMID 14517187
- [Background] Mancuso P, Rabascio C, Bertolini F. Strategies to investigate circulating endothelial cells in cancer. Pathophysiol Haemost Thromb. 2003 Sep-2004 Dec;33(5-6):503-6. doi: 10.1159/000083853. PMID 15692268
- [Background] Singh SK, Hawkins C, Clarke ID, Squire JA, Bayani J, Hide T, Henkelman RM, Cusimano MD, Dirks PB. Identification of human brain tumour initiating cells. Nature. 2004 Nov 18;432(7015):396-401. doi: 10.1038/nature03128. PMID 15549107